CLINICAL TRIAL: NCT05398757
Title: The Effect of Intraoperative Administration of Dexmedetomidine, Propofol and Midazolam on Postoperative Levels of Inflammatory Markers and Development of Postoperative Cognitive Dysfunction After Pertrochanteric Fracture Surgery.
Brief Title: Propofol and Dexmedetomidin vs Midazolam Intraoperative Sedation and POCD
Acronym: ProDex-POCD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too long recruitment period due to small number of patients
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OsijekPOCD
Record Dates: First submitted 2022-04-19; First posted 2022-06-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Pain, Acute; Pertrochanteric Fracture
Keywords: Postoperative Cognitive Dysfunction; Postoperative pain; Pertrochanteric Fracture; IL-6; Dexmedetomidin; Propofol; Midazolam; Sedation
MeSH Terms: conditions — Postoperative Cognitive Complications; Pain, Postoperative | interventions — Midazolam; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midazolam (Other): For sedation during surgery, patients will receive i.v. midazolam in dose 0.05 - 0.07 mg/kg.
  Interventions: Behavioral: Mini mental state exame (MMSE); Behavioral: Digit Symbol Substitution Test (DSST); Diagnostic Test: Numeric rating Scale (NRS); Diagnostic Test: Postoperative inflammation; Drug: Midazolam
- Propofol (Active Comparator): For sedation during surgery, patients will receive i.v. propofol in dose 25-27 mcg/kg/min.
  Interventions: Behavioral: Mini mental state exame (MMSE); Behavioral: Digit Symbol Substitution Test (DSST); Diagnostic Test: Numeric rating Scale (NRS); Diagnostic Test: Postoperative inflammation; Drug: Propofol
- Dexmedetomidin (Active Comparator): For sedation during surgery, patients will receive i.v. dexmedetomidin in dose 0.5 mcg/kg/h
  Interventions: Behavioral: Mini mental state exame (MMSE); Behavioral: Digit Symbol Substitution Test (DSST); Diagnostic Test: Numeric rating Scale (NRS); Diagnostic Test: Postoperative inflammation; Drug: Dexmedetomidin

INTERVENTIONS:
Behavioral: Mini mental state exame (MMSE) — Before the operation, and on the 1st, 3rd and 5th day after the operation, the Mini mental state exam (MMSE) score will be measured
Behavioral: Digit Symbol Substitution Test (DSST) — Before the operation, and on the 1st, 3rd and 5th day after the operation, the Digit Symbol Substitution Test (DSST) score will be measured
Diagnostic Test: Numeric rating Scale (NRS) — 4h, 8h, 12h and 24h after surgery, pain in all patients will be assessed by the NRS scale.
Diagnostic Test: Postoperative inflammation — All patients included in the study will have their blood taken for laboratory analysis of red blood cells, leukocytes, CRP, PCT, ChE and IL-6. Analyzes will be performed before the procedure, on the 1st, 3rd and 5th postoperative day.
Drug: Midazolam — For sedation during surgery, patients in midazolam group will receive i.v. midazolam in dose 0.05 - 0.07 mg/kg after spinal anesthesia.
  Other Names: Control - group M
  Arms: Midazolam
Drug: Propofol — For sedation during surgery, patients in propofol group will receive i.v. propofol in dose 25-27 mcg/kg/min.
  Other Names: Group P
  Arms: Propofol
Drug: Dexmedetomidin — For sedation during surgery, patients in dexmedetomidin gropu will receive i.v. dexmedetomidin in dose 0.5 mcg/kg/h
  Other Names: Group D
  Arms: Dexmedetomidin

SUMMARY:
This study will examine the effect of intraoperative sedation with midazolam, propofol and dexemdetomidine on the occurrence of postoperative cognitive impairment in patients undergoing surgical treatment of pertrochanteric fracture of the femur.

DETAILED DESCRIPTION:
Patients undergoing surgical treatment of pertrochanteric femoral fracture by intramedullary fixation will be included in the study. Patients will be older than 65 years and will belong to class I to III anesthesia risk according to the ASA classification. All patients included in the study will sign informed consent. Patients with dementia, mental illness, psychoorganically altered patients, and patients with a contraindication to dexmedetomidine, propofol, midazolam or with a contraindication to spinal anesthesia will be excluded from the study. All patients included in the study will have their blood taken for laboratory analysis of red blood cells, leukocytes, CRP, PCT, ChE and IL-6. Analyzes will be performed before the procedure, on the 1st, 3rd and 5th postoperative day. All patients will be tested for Mini mental state exame (MMSE) score before surgery to rule out pre-existing cognitive impairment, and those patients who have an MMSE value <17 prior to surgery will be excluded from the study. In premedication, patients will be randomized using three envelopes selected by the blind researcher for the contents of each envelope. According to envelope patients will be divided into three groups: dexmedetomidine group (DS), propofol group (PS) and midazolam group (MS). Neuroaxial spinal block with intrathecal administration of 12.5 - 15 mg 0.5% levobupivacaine in the intervertebral space L3 / L4 or L4 / L5 will be the technique of anesthesia. After spinal block, patients in the DS group will receive a continuous infusion of dexmedetomidine at a dose of 0.5 mcg / kg / h, patients in the PS group will receive a continuous infusion of propofol at a dose of 25-75 mcg / kg / min, while patients in the MS group will receive 0.05-0.07 mg / kg bolus i.v. midazolam. The total dose administered and the duration of surgery will be recorded. The volume of intraoperatively administered crystalloids or blood products will be recorded in all patients included in the study. In the postoperative period, pain will be measured with a numerical rating scale (NRS) 4, 8, 12 and 24 hours after surgery. All patients will receive the usual postoperative analgesia with metamizole and tramadol according to the protocol of the Department. On the 1st, 3rd and 5th postoperative days in the morning between 8.00 and 10.00, all patients will be tested for MMSE and Digit Symbol Substitution Test (DSST) score. A researcher who will evaluate MMSE and DSST values in the postoperative period will be blind to the drug that patients received intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Pertrochanteric fracture surgery
* Informed consent signed

Exclusion Criteria:

* MMSE before surgery < 17
* Allergy on midazolam, propofol or dexemdetomidine
* Contraindication for neuroaxial anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of postoperative cognitive dysfunction (POCD) measured by MMSE | 5 days
  The incidence of POCD with respect to intraoperative sedation in the postoperative period will be measured by MMSE test on the first, third and fifth postoperative day. An absolute z-score greater than 1.96 in postoperative testing or a decrease in the postoperative MMSE value by more than 20% relative to the preoperative value will be considered the occurrence of POCD in the postoperative period.
Occurrence of postoperative cognitive dysfunction (POCD) measured by DSST | 5 days
  The incidence of POCD with respect to intraoperative sedation in the postoperative period will be measured by DSST on the first, third and fifth postoperative day. An absolute z-score greater than 1.96 in postoperative testing or a decrease in the postoperative DSST value by more than 20% relative to the preoperative value will be considered the occurrence of POCD in the postoperative period.
Postoperative inflammation measured by serum CRP levels | 5 days
  Postoperative inflammation with respect to intraoperative sedation will be assessed by serum levels of CRP at postoperative day 1, 3 and 5. CRP > 50 mg/L and rising dynamic of CRP in postoperative serial measurements will be considered as systemic inflammation state.
Postoperative inflammation measured by white blood cells count | 5 days
  Postoperative inflammation with respect to intraoperative sedation will be assessed by serum levels of white blood cells. Leukocytes > 12.000/mm3 or < 4.000/mm3 in postoperative serial measurements will be considered as systemic inflammation state.
Postoperative inflammation measured by serum IL-6 levels | 5 days
  Postoperative inflammation with respect to intraoperative sedation will be assessed by serum levels IL-6 at postoperative day 1, 3 and 5. Continuous increase of IL-6 in postoperative serial measurements will be considered as systemic inflammation state.
Postoperative inflammation measured by serum cholinesterase activity | 5 days
  Postoperative inflammation with respect to intraoperative sedation will be assessed by serum cholinesterase activity at postoperative day 1, 3 and 5. Cholinesterase activity < 4000 U/L in postoperative serial measurements will be considered as systemic inflammation state.
Postoperative inflammation measured by serum PCT levels | 5 days
  Postoperative inflammation with respect to intraoperative sedation will be assessed by serum levels of PCT at postoperative day 1, 3 and 5. PCT > 0.5 ng/ml and continuous increase in postoperative serial measurements will be considered as systemic inflammation state.

SECONDARY OUTCOMES:
Postoperative pain | 24 hours
  Postoperative pain with respect to intraoperative sedation will be examined by Numeric rating scale (NRS) 4, 8, 12 and 24 hours after surgery. NRS is a scale from 0 to 10, where 0 means no pain and 10 means the strongest pain. NRS above or equal to 4 will be considered inadequate postoperative analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Nenad Neskovic, PhD, Principal Investigator — University Hospital Osijek
Locations (1):
- University Hospital Osijek, Osijek, Croatia

REFERENCES:
- [Background] Monk TG, Price CC. Postoperative cognitive disorders. Curr Opin Crit Care. 2011 Aug;17(4):376-81. doi: 10.1097/MCC.0b013e328348bece. PMID 21716111
- [Background] Urits I, Orhurhu V, Jones M, Hoyt D, Seats A, Viswanath O. Current Perspectives on Postoperative Cognitive Dysfunction in the Ageing Population. Turk J Anaesthesiol Reanim. 2019 Dec;47(6):439-447. doi: 10.5152/TJAR.2019.75299. Epub 2019 Sep 2. PMID 31828240
- [Background] Xiao QX, Liu Q, Deng R, Gao ZW, Zhang Y. Postoperative cognitive dysfunction in elderly patients undergoing hip arthroplasty. Psychogeriatrics. 2020 Jul;20(4):501-509. doi: 10.1111/psyg.12516. Epub 2020 Jan 24. PMID 31976614
- [Background] Rasmussen LS, Larsen K, Houx P, Skovgaard LT, Hanning CD, Moller JT; ISPOCD group. The International Study of Postoperative Cognitive Dysfunction. The assessment of postoperative cognitive function. Acta Anaesthesiol Scand. 2001 Mar;45(3):275-89. doi: 10.1034/j.1399-6576.2001.045003275.x. PMID 11207462
- [Background] Tombaugh TN, McIntyre NJ. The mini-mental state examination: a comprehensive review. J Am Geriatr Soc. 1992 Sep;40(9):922-35. doi: 10.1111/j.1532-5415.1992.tb01992.x. PMID 1512391
- [Background] van Sinderen K, Schwarte LA, Schober P. Diagnostic Criteria of Postoperative Cognitive Dysfunction: A Focused Systematic Review. Anesthesiol Res Pract. 2020 Nov 16;2020:7384394. doi: 10.1155/2020/7384394. eCollection 2020. PMID 33281900
- [Background] Wang K, Wu M, Xu J, Wu C, Zhang B, Wang G, Ma D. Effects of dexmedetomidine on perioperative stress, inflammation, and immune function: systematic review and meta-analysis. Br J Anaesth. 2019 Dec;123(6):777-794. doi: 10.1016/j.bja.2019.07.027. Epub 2019 Oct 24. PMID 31668347
- [Background] Mei B, Li J, Zuo Z. Dexmedetomidine attenuates sepsis-associated inflammation and encephalopathy via central alpha2A adrenoceptor. Brain Behav Immun. 2021 Jan;91:296-314. doi: 10.1016/j.bbi.2020.10.008. Epub 2020 Oct 8. PMID 33039659
- [Background] Hohener D, Blumenthal S, Borgeat A. Sedation and regional anaesthesia in the adult patient. Br J Anaesth. 2008 Jan;100(1):8-16. doi: 10.1093/bja/aem342. PMID 18070783
- [Background] Tobias JD, Leder M. Procedural sedation: A review of sedative agents, monitoring, and management of complications. Saudi J Anaesth. 2011 Oct;5(4):395-410. doi: 10.4103/1658-354X.87270. PMID 22144928
- [Background] Chen RM, Chen TG, Chen TL, Lin LL, Chang CC, Chang HC, Wu CH. Anti-inflammatory and antioxidative effects of propofol on lipopolysaccharide-activated macrophages. Ann N Y Acad Sci. 2005 May;1042:262-71. doi: 10.1196/annals.1338.030. PMID 15965071
- [Background] Kochiyama T, Li X, Nakayama H, Kage M, Yamane Y, Takamori K, Iwabuchi K, Inada E. Effect of Propofol on the Production of Inflammatory Cytokines by Human Polarized Macrophages. Mediators Inflamm. 2019 Mar 17;2019:1919538. doi: 10.1155/2019/1919538. eCollection 2019. PMID 31007601